CLINICAL TRIAL: NCT06792032
Title: The Effect of Peer Mentoring Model Supported by Mobile Application on Individual, Social, and Academic Success of Nursing Students
Brief Title: The Effect of Peer Mentoring Model Supported by Mobile Application
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Seda Tugba Baykara Mat, Asst. Prof., University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: The Effect of Peer Mentoring
Record Dates: First submitted 2024-12-04; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Peer Group Guidance; Academic Achievements; Nursing; Mobile Applications; College Adaptation; Self Efficacy; Mentoring
Keywords: Mobile Applications; Academic Achievement; Peer Group Guidance; College Adaptation; Self Efficacy

STUDY DESIGN:
Intervention Model Description: Study Design: This study is designed as a randomized controlled experimental study to assess the impact of a peer guidance model supported by a mobile application on the individual, social, and academic success of nursing students.
  Dependent Variables:
  Individual success: self-efficacy levels Social success: university adaptation levels Academic success: satisfaction with education and academic achievement Independent Variable: The peer guidance model supported by the mobile application.
  Location of the Study: The study will be conducted at the Nursing Department of a Faculty of Health Sciences in Istanbul, with participation from students attending clinical courses.
  Population and Sample:
  The population of the study consists of approximately 306 nursing students enrolled in the Nursing Department between September 2024 and June 2025. The study aims to include the entire population without using any sampling method. The plan is for 3rd and 4th-year students to act as peer guides (m
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer mentoring model supported by mobile application (Experimental): Population and Sample:
  The study population consists of approximately 306 nursing students enrolled in the Nursing Department between September 2024 and June 2025. It aims to include the entire population without using any sampling method. The plan is for third -and fourth-year students to act as peer guides (mentors), while first -and second-year students will be mentees.
  1st and 2nd-year students: 85+80 = 165 3rd and 4th-year students: 70+71 = 141 Additionally, 4th-year students will be assigned as peer guides for 1st-year students. In a similar study by Cant and Cooper (2017), the effect size was calculated as 0.80. Based on power analysis, to achieve a 95% power, with a 5% significance level and an effect size of 0.80, a sample size of 70 (35 experimental and 35 control group) is required (df=68; t=1.667). Considering the test's high power and potential dropouts, the study aims to recruit 90 participants (45 per group).Peer mentoring model supported by mobile application
  Interventions: Other: peer mentoring with mobile application
- 2. group nursing students (No Intervention): Nursing students with no intervention

INTERVENTIONS:
Other: peer mentoring with mobile application — peer mentoring with mobile application
  Arms: Peer mentoring model supported by mobile application

SUMMARY:
This study investigates the effects of a peer-guided model supported by a mobile application on nursing students' educational processes. The primary goal of the research is to assess the potential impact of this model on students' self-efficacy, university adaptation, and academic success.

The study will be conducted as a randomized controlled experimental design with 70 nursing students. The experimental group will have 35 students, while the control group will also include 35 students. The data collection tools will include a student diagnostic form, university adaptation scale, satisfaction with educational methods scale, academic self-efficacy scale, and academic achievement scale.

The research process will include the application of the student diagnostic form, the development of the mobile application, an informational meeting about the peer-guided model for students, randomization, mentor-mentee assignments, initial data collection, and the stages of initiation, training, separation, and re-evaluation. The use of the peer guidance model and mobile application will be emphasized during the educational process. Motivating peer leaders and achieving the program's objectives will be ensured through peer leader seminars.

Data analysis will be performed using SPSS 25.0 software, with an initial examination of the data distribution. T-tests or one-way ANOVA will be used for normally distributed variables, and the Scheffe test will be applied to identify differences. Mann-Whitney U and Kruskal-Wallis tests will be used for non-normally distributed variables. Additionally, Pearson correlation analysis will determine relationships between continuous variables. The effects of independent variables will be evaluated using multiple regression analysis (Backward method). Statistical significance will be assessed at a p-value of <0.05.

This study has been designed according to CONSORT standards, and all necessary ethical approvals and institutional permissions have been obtained.

DETAILED DESCRIPTION:
The project contributes to the knowledge base by bridging the gap between nursing education and mobile technology. While there is limited research in the literature on the impact of peer-guided models and mobile applications compared to traditional teaching methods, this project aims to address this knowledge gap. It will explore how such a model can enhance the educational experience of nursing students and contribute to their professional development.

The proposed new technology and method will offer various contributions to the literature:

Mobile Application:

The mobile application, designed to focus on the professional development of nursing students, will offer a unique feature that enables students to engage in interactive learning environments through the peer-guided model in a novel way. The application will be significant for its unique interface and personalized recommendations tailored to the students' needs. Additionally, designing the application specifically for nursing students positions it uniquely within its target audience, while its capacity for developing new modules and adaptability to technological innovations strengthens its applicability for other student groups in different professions. These elements will help position the application competitively in the long term, offering a potential competitive edge.

Practical Application Opportunity:

This project enables nursing students to combine theoretical knowledge with practical applications, thereby enhancing their professional skills. It provides a new perspective on the integration of mobile technology into educational practices, emphasizing the importance of this fusion in fostering practical experience for students, as suggested by current literature.

Improvement of the Learning Experience:

The use of the peer-guided model and mobile application will increase interaction among students, enriching their learning experiences. This represents a new approach to providing support and collaboration opportunities that are often absent in traditional classroom settings.

Evaluation of Technology-Supported Peer Guidance Model:

The value of this project lies in its systematic evaluation of how the peer-guided model in education can be enhanced through the use of a mobile application, and its subsequent effects on students' academic success, self-efficacy, and satisfaction.

Exploration of Innovative Educational Approaches:

This study investigates how technology can be integrated into the learning process, differing from traditional educational approaches. By examining the effects of a mobile application-supported peer-guided model on student performance and experiences, the research will offer a fresh perspective in the literature.

Development of Student-Centered Learning Environments:

The mobile application proposed in the project will provide tools that allow students to actively manage their learning processes. This will represent a significant step in creating student-centered learning environments and contribute to the literature on student autonomy in learning.

New Technology, Methods, and Theories:

The mobile application-supported peer guidance model presents an innovative approach, different from traditional peer guidance practices. By combining peer support with the power of mobile technology, it aims to provide a more effective learning experience for students.

Thus, the new technology and method proposed in this project will provide a fresh perspective and application framework for peer-guided models in education, offering valuable contributions to the literature on nursing education.

Hypotheses:

* H1: The mobile application-supported peer guidance model has an impact on nursing students' university adaptation process.
* H2: The mobile application-supported peer guidance model affects nursing students' academic self-efficacy levels.
* H3: The mobile application-supported peer guidance model has an effect on nursing students' academic success.
* H4: The mobile application-supported peer guidance model impacts nursing students' satisfaction with teaching methods.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* To be enrolled in the Department of Nursing
* Continuing formal education
* Internet access
* Using a smart phone

Exclusion Criteria:

* Enrolled in a different programme
* Department/school change
* The student's desire to leave the study

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
Academic Success, Self-efficacy Level, Satisfaction Surveys: | "up to 12 months"
  Academic Success: The mobile application used within the scope of the project is expected to improve the academic performance of the students.
  whether it improves or not can be measured. Students' course grades, exam performance and general academic achievement can be taken into consideration.
  can be evaluated by taking into consideration. Self-efficacy Level: Increased self-efficacy of nursing students through mobile application and peer mentoring programme.
  self-efficacy levels can be measured. Students' level of self-confidence, problem solving skills and s elf-efficacy can be measured.
  Their ability to make decisions on their own can be assessed. Satisfaction Surveys: Regular satisfaction surveys to nursing students during the project process the extent to which they were satisfied with the mobile application and peer mentoring programme and what kind of improvements can be identified that they want

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Beykent University, Istanbul, Büyükçekmece
  - Istanbul Beykent University, Istanbul

IPD SHARING:
Plan to Share IPD: No
IPD is typically not shared in order to protect participants' privacy and comply with ethical and legal regulations.